CLINICAL TRIAL: NCT01185262
Title: Phase I Study of the Activity and Safety of Lenalidomide and Rituximab as Non-chemotherapy Therapy for Patients With Recurrent and Refractory Chronic Lymphocytic Leukemia
Brief Title: Activity & Safety Study of Lenalidomide & Rituximab as Non-chemotherapy Based Therapy on Chronic Lymphocytic Leukemia
Acronym: LLC-LENAR-08
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MD Anderson International Spain SA (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LLC-LENAR-08; LLC-LENAR-08 (Other: Fundación MD Anderson Internacional. España); NCT01348815 (obsolete NCT alias)
Record Dates: First submitted 2009-12-17; First posted 2010-08-19 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Recurrent and refractory chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomida, Rituximab (Experimental): Phase I: Lenalidomide will be administered from day 1 to 21 of 28 days cycles, escalating doses (from 2,5mg to 25 mg).Rituximab dose will be administered at the standard (375 mg/m2 in the first cycle and 500 mg/m2 in successive cycles).
  Interventions: Drug: Lenalidomida and Rituximab

INTERVENTIONS:
Drug: Lenalidomida and Rituximab — Lenalidomide: Oral use. It will be administered from day 1 to 21 of 28 days cycles in a total of 6 cycles.
  Rituximab, intravenous use. The dose will be administered at the standard (375 mg/m2 in the first cycle and 500 mg/m2 in successive cycles).
  In the first cycle Rituximab will be administered in two divided doses:100mg/m2 total on day 1 and the rest up to 375mg/m2 on day 2.
  If lenalidomide treatment starts on day 1, Rituximab will be administered, in this first cycle, on days -2 (100 mg/m2) and -1 (275 mg/m2).
  In the second and subsequent cycles, 500 mg/m2 of Rituximab will be administered on day -1.
  Other Names: Lenalidomide: REVLIMID; Rituximab: MABTHERA

SUMMARY:
The rationale for combining lenalidomide with rituximab derives from preclinical observations suggesting that lenalidomide may enhance the ADCC (antigen-dependent cellular cytotoxicity) triggered by monoclonal antibodies such as rituximab. Lenalidomide augments NK cytotoxicity by increasing CD56dimCD3 subset, in addition to inducing IL-2 in T cells. These results provide the cellular and molecular basis for the use of lenalidomide as an adjuvant in immunotherapeutic strategies of monoclonal antibodies (mAb)-based therapies. The combination lenalidomide-rituximab was tested in lymphoma cell lines but not specifically on CLL cell lines. However the observed synergism was attributed to NK cells expansion, thus lending support to the notion that this synergism may operate in other B-cell lymphoproliferative malignancies.

The objective was to develop a non-cytotoxic and effective treatment for CLL that would fulfill an unmet medical need, as a significant proportion of CLL patients are elderly and frail. These patients experience an excess in chemotherapy induced toxicity, often preventing the completion of the planned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent and refractory CLL patients that have received at least one previous treatment with purine analogs.
* Adequate liver function and renal function.
* ECOG performance status ≤ 2.
* Signed informed consent
* Male and female patients who are fertile agree to use an effective barrier method of birth control to avoid pregnancy.

Exclusion Criteria:

* Positive serological markers for hepatitis B with the exception of HBsAc in previously vaccinated patients
* Pregnant patients
* HIV infection
* Concurrent chemotherapy or immunotherapy
* Other malignancy within the last 2 years, except for localized cutaneous carcinoma
* Neurological impairment precluding understanding of protocol and the entailed visits and procedures.
* Patients with Renal insufficiency that requires dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-04; Primary Completion 2012-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Phase I: To determine Starting Recommended Dose for the first cycle and the subsequent cycles (Maximal Tolerated Dose)in relapsed B-cell CLL patients. | 5 months
  6 treatment cycles followed by an evaluation visit (between 60-90 days after last dosing) and quarterly follow up visits, until disease progression. Module I: patients on every cohort will have the same dose during treatment, except if they experiment DLT, in which case dose will be decreased (unless they are on the first dose level).

SECONDARY OUTCOMES:
To determine the toxicity profile of LenRtx. | 5 months
  Phase II: patients will be followed during 6 cycles, safety assessment visit and quarterly follow up visits
To determine the time to treatment failure. | 5 months
  Phase II: patients will be followed during 6 cycles, safety assessment visit and quarterly follow up visits
To determine the molecular response rate. | 5 months
  Phase II: patients will be followed during 6 cycles, safety assessment visit and quarterly follow up visits
To determine the clinical response rate (combined morphological and flow cytometry criteria). | 5 months
  6 treatment cycles followed by an evaluation visit (between 60-90 days after last dosing) and quarterly follow up visits, until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: José F Tomas, MD, Principal Investigator — MD Anderson Internacional España
Locations (7):
- Spain (7):
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - MD Anderson Internacional España, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Clínico de Salamanca, Salamanca, Salamanca
  - Hospital Virgen del Rocío, Seville, Sevilla
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza